CLINICAL TRIAL: NCT07371247
Title: Based on ctDNA-MRD Guided Adjuvant Treatment Escalation After Definitive Chemoradiotherapy for Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma: a Study on Safety and Efficacy
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-1071
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer; MRD; ctDNA
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD-positive groups (Active Comparator): Assessed as MRD-positive based on ctDNA testing
  Interventions: Drug: Step-up therapy
- MRD-negative groups (Sham Comparator): Assessed as MRD-negative based on ctDNA testing
  Interventions: Drug: Standard treatment Routine treatment

INTERVENTIONS:
Drug: Step-up therapy — Patients receive step-up therapy, consisting of 4 cycles of immunotherapy combined with intravenous chemotherapy, followed by immunotherapy plus oral chemotherapy for 6 months. MRD testing is repeated after the completion of immunotherapy combined with intravenous chemotherapy.
  Arms: MRD-positive groups
Drug: Standard treatment Routine treatment — Patients receive 2 cycles of consolidative intravenous chemotherapy and then proceed to routine follow-up. MRD testing is repeated after the completion of chemotherapy.
  Arms: MRD-negative groups

SUMMARY:
Numerous studies have confirmed that ctDNA-MRD detection technology based on peripheral blood can identify minimal residual disease (MRD) following surgery and other curative treatments, indicating a higher risk of recurrence. Multiple exploratory studies in esophageal cancer have demonstrated that patients who are ctDNA-MRD positive after definitive chemoradiotherapy (dCRT) exhibit poorer progression-free survival (PFS) and a higher risk of recurrence. Furthermore, the recent NEXUS-1 translational study confirmed that 66.7% of unresectable patients achieved the goal of conversion surgery after receiving definitive chemoradiotherapy combined with immunotherapy. Notably, patients who were ctDNA-MRD positive after chemoradiotherapy had a significantly worse prognosis. These findings suggest that ctDNA-MRD status after chemoradiotherapy has prognostic stratification value and that consolidative immunotherapy is effective.

Based on these previous discoveries, this study aims to investigate the safety and efficacy of an escalated treatment strategy involving immunotherapy combined with chemotherapy for high-risk populations after definitive chemoradiotherapy for esophageal cancer, guided by personalized MRD detection results.

ELIGIBILITY:
* Inclusion Criteria

  1. Histologically confirmed locally advanced esophageal squamous cell carcinoma (ESCC), with clinical stage Ⅱ-Ⅳ unresectable disease (including unresectable cases, patients with surgical contraindications, or those who refuse surgery). According to the 8th edition AJCC staging system, the pretreatment clinical stage is defined as: cT1N2-3M0, cT2-4bN0-3M0; M1 disease is limited to non-regional lymph node metastases, excluding distant organ metastases.
  2. No prior systemic therapy administered for the disease, and planned to receive definitive chemoradiotherapy (dCRT).
  3. Having undergone 1021-gene large panel testing on tissue samples.
  4. Aged 18-80 years old.
  5. Expected overall survival ≥ 6 months.
  6. ECOG performance status 0-1.
  7. Normal blood biochemical parameters, with normal liver and kidney function.
  8. Able to understand the study protocol, voluntarily participate in the study, and sign the informed consent form.
  9. Good compliance, able to cooperate with specimen collection at all designated time points and provide relevant clinical data.
* Exclusion Criteria

  1. Have participated in other clinical trials within 3 months prior to enrollment.
  2. Have a history of other malignant tumors within 3 years prior to the diagnosis of esophageal cancer.
  3. Have a history of severe mental illness.
  4. Patients who are unable to understand the study protocol and thus cannot cooperate, or who refuse to sign the informed consent form.
  5. Have contraindications to chemoradiotherapy.
  6. Have a history of autoimmune diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen B, Liu S, Zhu Y, Wang R, Cheng X, Chen B, Dragomir MP, Zhang Y, Hu Y, Liu M, Li Q, Yang H, Xi M. Predictive role of ctDNA in esophageal squamous cell carcinoma receiving definitive chemoradiotherapy combined with toripalimab. Nat Commun. 2024 Mar 1;15(1):1919. doi: 10.1038/s41467-024-46307-7. PMID 38429311
- [Result] Takei S, Kotani D, Laliotis G, Sato K, Fujiwara N, Kawazoe A, Hashimoto T, Mishima S, Nakayama I, Nakamura Y, Bando H, Kuboki Y, Sakashita S, Spickard E, George GV, Dutta P, Sharma S, Malhotra M, Sethi H, Jurdi A, Liu MC, Yoshino T, Shitara K, Kojima T, Fujita T. Circulating Tumor DNA Assessment to Predict Risk of Recurrence after Surgery in Patients with Locally Advanced Esophageal Squamous Cell Carcinoma: A Prospective Observational Study. Ann Surg. 2025 Mar 21. doi: 10.1097/SLA.0000000000006699. Online ahead of print. PMID 40115982
- [Result] Liu Z, Wang G, Yang Y, Su Y, Zhang H, Liu J, Cui P, Fan X, Yang J, Zhang Z, Gao X, Chao Y, Mostert B, van Lanschot JJB, Wijnhoven BPL, Law S, Li C, Cai S, Li Z. ctDNA detects residual disease after neoadjuvant chemoradiotherapy and guides adjuvant therapy in esophageal squamous cell carcinoma. Cell Rep Med. 2025 Sep 16;6(9):102334. doi: 10.1016/j.xcrm.2025.102334. Epub 2025 Sep 5. PMID 40914168
- [Result] Driessen RS, van Diemen PA, Raijmakers PG, Knuuti J, Maaniitty T, Underwood SR, Nagel E, Robbers LFHJ, Demirkiran A, von Bartheld MB, van de Ven PM, Hofstra L, Somsen GA, Tulevski II, Boellaard R, van Rossum AC, Danad I, Knaapen P. Functional stress imaging to predict abnormal coronary fractional flow reserve: the PACIFIC 2 study. Eur Heart J. 2022 Sep 1;43(33):3118-3128. doi: 10.1093/eurheartj/ehac286. PMID 35708168
- [Result] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Result] Ajani JA, D'Amico TA, Almhanna K, Bentrem DJ, Besh S, Chao J, Das P, Denlinger C, Fanta P, Fuchs CS, Gerdes H, Glasgow RE, Hayman JA, Hochwald S, Hofstetter WL, Ilson DH, Jaroszewski D, Jasperson K, Keswani RN, Kleinberg LR, Korn WM, Leong S, Lockhart AC, Mulcahy MF, Orringer MB, Posey JA, Poultsides GA, Sasson AR, Scott WJ, Strong VE, Varghese TK Jr, Washington MK, Willett CG, Wright CD, Zelman D, McMillian N, Sundar H; National comprehensive cancer network. Esophageal and esophagogastric junction cancers, version 1.2015. J Natl Compr Canc Netw. 2015 Feb;13(2):194-227. doi: 10.6004/jnccn.2015.0028. PMID 25691612
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338